CLINICAL TRIAL: NCT01702636
Title: STOP-AUST: The Spot Sign and Tranexamic Acid On Preventing ICH Growth - AUStralasia Trial.
Acronym: STOP-AUST
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Neuroscience Trials Australia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NTA1201
Record Dates: First submitted 2012-10-03; First posted 2012-10-08 (Estimated); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Intracerebral Haemorrhage; Stroke
Keywords: Intracerebral Hemorrhage; ICH; Stroke; Cerebrovascular Disorders; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Vascular Diseases; Cardiovascular Diseases; Tranexamic Acid; Antifibrinolytic Agents; Fibrin Modulating Agents; Pharmacologic Actions; Cardiovascular Agents; Therapeutic Uses; Hematologic Agents; Hemostatics; Contrast Media; Angiography; Cerebral Angiography; Tomography, X-Ray Computed
MeSH Terms: conditions — Cerebral Hemorrhage; Stroke; Cerebrovascular Disorders; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Vascular Diseases; Cardiovascular Diseases | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tranexamic Acid (Active Comparator): Intravenous tranexamic acid 1000 mg in 100 mL 0.9% NaCl over 10 minutes followed by 1000 mg in 500 mL 0.9% NaCl infusion over 8 hours.
  Interventions: Drug: Tranexamic Acid
- Placebo (Placebo Comparator): Intravenous placebo in 100 mL 0.9% NaCl over 10 minutes followed by 500 mL 0.9% NaCl infusion over 8 hours.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tranexamic Acid
  Arms: Tranexamic Acid
Drug: Placebo
  Arms: Placebo

SUMMARY:
The aim of the study is to test if intracerebral haemorrhage (ICH) patients who have contrast extravasation on computed tomography angiography, the "spot sign", have lower rates of haematoma growth when treated with tranexamic acid within 4.5 hours of stroke onset, compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with an acute ICH
* Contrast extravasation within the haemorrhage, "spot sign", evaluated from the CTA according to three criteria, all of which must be present:

  1. Serpiginous or spot-like appearance within the margin of a parenchymal haematoma without connection to an outside vessel;
  2. The density (in Hounsfield units) should be greater than that of the background haematoma (site investigators are not required to document the density); and
  3. No hyperdensity at the corresponding location on non-contrast CT.
* Age ≥18 years
* Treatment can commence within 1 hour of initial CT and within 4.5 hours of symptom onset (or in patients with unknown time of symptom onset, the time patient was last known to be well)
* Informed consent has been received in accordance to local ethics committee requirements

Exclusion Criteria:

* Glasgow coma scale (GCS) total score of <8
* Brainstem ICH
* ICH volume >70 ml as measured by the ABC/2 method
* ICH known or suspected by study investigator to be secondary to trauma, aneurysm, vascular malformation, haemorrhagic transformation of ischaemic stroke, cerebral venous thrombosis, thrombolytic therapy, tumor, or infection
* Contrast already administered within 24 hours prior to initial CT or contraindication to imaging with CT contrast agents (e.g. known or suspected iodine allergy or significant renal failure)
* Any history or current evidence suggestive of venous or arterial thrombotic events within the previous 12 months, including clinical, ECG, laboratory, or imaging findings. Clinically silent chance findings of old ischemia are not considered exclusion.
* Hereditary or acquired haemorrhagic diathesis or coagulation factor deficiency.
* Use of heparin, low-molecular weight heparin, GPIIb/IIIa antagonist, or oral anticoagulation (e.g. warfarin, factor Xa inhibitor, thrombin inhibitor) within the previous 14 days, irrespective of laboratory values
* Pregnancy (women of childbearing potential must be tested)
* Planned surgery for ICH within 24 hours
* Concurrent or planned treatment with haemostatic agents (e.g. prothrombin complex concentrate, vitamin K, fresh frozen plasma, or platelet transfusion)
* Participation in any investigational study in the last 30 days
* Known terminal illness or planned withdrawal of care or comfort care measures.
* Any condition that, in the judgment of the investigator could impose hazards to the patient if study therapy is initiated or affect the participation of the patient in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-12 (Actual); Primary Completion 2019-08-14 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
ICH growth by 24±3 hours as defined by either 33% or 6 ml increase from baseline, adjusted for baseline ICH volume. | 24+/-3 hours

SECONDARY OUTCOMES:
Major thromboembolic events (myocardial infarction, ischaemic stroke, pulmonary embolism) | Within 90+/-7 days
Absolute ICH growth volume by 24±3 hours, adjusted for baseline ICH volume | 24+/-3 hours
Absolute intraventricular haematoma (IVH) growth volume by 24±3 hours, adjusted for baseline IVH volume | 24+/-3 hours
modified Rankin Scale (mRS) score of 0-4 at 3 months | 90+/-7 days
modified Rankin Scale (mRS) score of 0-3 at 3 months | 90+/-7 days
Categorical shift in mRS at 3 months, subject to the validity of proportional odds assumption | 90+/-7 days
Death due to any cause by 3 months | within 90+/-7 days

OTHER OUTCOMES:
ICH growth | 24+/-3 hours
  Exploratory analyses will be run with adjustments for baseline variables such as age, Glasgow Coma Scale (GCS), presence of IVH, and ICH location, and in the following subgroups: onset-to-treatment time (<3 vs. >3 hours); baseline ICH volume (<30 vs. >30 ml); anatomical location (deep, lobar, or cerebellar); IVH (absent vs. present); GCS (>12 vs. 8-12) and age (<70 vs. >70). These analyses will be hypothesis generating, as the trial is not powered for them.
modified Rankin Scale (mRS) | 90+/-7 days
  Exploratory analyses will be run with adjustments for baseline variables such as age, Glasgow Coma Scale (GCS), presence of IVH, and ICH location, and in the following subgroups: onset-to-treatment time (<3 vs. >3 hours); baseline ICH volume (<30 vs. >30 ml); anatomical location (deep, lobar, or cerebellar); IVH (absent vs. present); GCS (>12 vs. 8-12) and age (<70 vs. >70). These analyses will be hypothesis generating, as the trial is not powered for them.

CONTACTS AND LOCATIONS:
Overall Officials: Atte Meretoja, MD, Principal Investigator — The Florey Institute of Neuroscience and Mental Health; Geoffrey A Donnan, MD, Principal Investigator — The Florey Institute of Neuroscience and Mental Health; Stephen M Davis, MD, Principal Investigator — Melbourne Health
Locations (11):
- Australia (10):
  - Gosford Hospital, Kanwal, New South Wales
  - John Hunter Hospital, Newcastle, New South Wales
  - St. Vincent's Hospital, Sydney, New South Wales
  - Royal Prince Alfred Hospital, Sydney, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Box Hill Hospital, Box Hill, Victoria
  - Western Hospital, Footscray, Victoria
  - Frankston Hospital, Frankston, Victoria
  - The Royal Melbourne Hospital, Melbourne, Victoria
- Helsinki University Central Hospital, Helsinki, Finland

REFERENCES:
- [Derived] Eilertsen H, Menon CS, Law ZK, Chen C, Bath PM, Steiner T, Desborough MJ, Sandset EC, Sprigg N, Al-Shahi Salman R. Haemostatic therapies for stroke due to acute, spontaneous intracerebral haemorrhage. Cochrane Database Syst Rev. 2023 Oct 23;10(10):CD005951. doi: 10.1002/14651858.CD005951.pub5. PMID 37870112
- [Derived] Yogendrakumar V, Wu TY, Churilov L, Tatlisumak T, Strbian D, Jeng JS, Kleinig TJ, Sharma G, Campbell BC, Zhao H, Hsu CY, Meretoja A, Donnan GA, Davis SM, Yassi N. Does tranexamic acid affect intraventricular hemorrhage growth in acute ICH? An analysis of the STOP-AUST trial. Eur Stroke J. 2022 Mar;7(1):15-19. doi: 10.1177/23969873211072402. Epub 2022 Feb 1. PMID 35300248
- [Derived] Meretoja A, Yassi N, Wu TY, Churilov L, Sibolt G, Jeng JS, Kleinig T, Spratt NJ, Thijs V, Wijeratne T, Cho DY, Shah D, Cloud GC, Phan T, Bladin C, Moey A, Aviv RI, Barras CD, Sharma G, Hsu CY, Ma H, Campbell BCV, Mitchell P, Yan B, Parsons MW, Tiainen M, Curtze S, Strbian D, Tang SC, Harvey J, Levi C, Donnan GA, Davis SM. Tranexamic acid in patients with intracerebral haemorrhage (STOP-AUST): a multicentre, randomised, placebo-controlled, phase 2 trial. Lancet Neurol. 2020 Dec;19(12):980-987. doi: 10.1016/S1474-4422(20)30369-0. Epub 2020 Oct 28. PMID 33128912
- [Derived] Meretoja A, Churilov L, Campbell BC, Aviv RI, Yassi N, Barras C, Mitchell P, Yan B, Nandurkar H, Bladin C, Wijeratne T, Spratt NJ, Jannes J, Sturm J, Rupasinghe J, Zavala J, Lee A, Kleinig T, Markus R, Delcourt C, Mahant N, Parsons MW, Levi C, Anderson CS, Donnan GA, Davis SM. The spot sign and tranexamic acid on preventing ICH growth--AUStralasia Trial (STOP-AUST): protocol of a phase II randomized, placebo-controlled, double-blind, multicenter trial. Int J Stroke. 2014 Jun;9(4):519-24. doi: 10.1111/ijs.12132. Epub 2013 Aug 26. PMID 23981692